CLINICAL TRIAL: NCT02464397
Title: A Randomized Prospective Multicenter Trial to Examine Vascular Healing at 1 and 6 Month(s) After Deployment of TItanium-nitride-oxide-coated OPTIMAX™ Bio-active-stent (BAS) Stent and SYNERGY™ Everolimus-Eluting Stent (EES) in Patients With Acute Coronary Syndromes by Means of Optical Coherence Tomography
Brief Title: Comparison of Strut Coverage With OPTIMAX Versus SYNERGY Stents
Acronym: OPTIMAX-OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Principal Investigator, Pasi Karjalainen, Professor, The Hospital District of Satakunta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA-010
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Vascular healing of coronary stents in patients with acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OPTIMAX-BAS 1 (Experimental): Titanium-nitride-oxide coated cobalt-chromium OPTIMAX™ bio-active stent (BAS). Patients will have OCT follow-up 1 month after the index procedure.
  Interventions: Device: Stent
- SYNERGY-EES 1 (Active Comparator): SYNERGY™ everolimus eluting stent (EES). Patients will have OCT follow-up 1 month after the index procedure.
  Interventions: Device: Stent
- OPTIMAX-OCT 6 (Experimental): Titanium-nitride-oxide coated cobalt-chromium OPTIMAX™ bio-active stent (BAS). Patients will have OCT follow-up 6 months after the index procedure.
  Interventions: Device: Stent
- SYNERGY-EES 6 (Active Comparator): SYNERGY™ everolimus eluting stent (EES). Patients will have OCT follow-up 6 months after the index procedure.
  Interventions: Device: Stent

INTERVENTIONS:
Device: Stent — In the study, either OPTIMAX or SYNERGY stent will be implanted in coronary artery lesion
  Other Names: PCI

SUMMARY:
The purpose of this study is to compare vascular healing of the stented segment after deployment of titanium-nitride-oxide coated cobalt-chromium OPTIMAX™ bio-active stent (BAS) and SYNERGY™ everolimus-eluting stent (EES) in patients with acute coronary syndromes requiring percutaneous coronary intervention.

Patients treated with BAS will be treated with DAPT for at least 4 weeks after the procedure followed by aspirin alone, while patients in the EES group will be treated with DAPT, at least for 6 months post procedure. In addition, this study will collect initial information about the safety and effectiveness of the BAS in comparison with EES group at 30 days, 6 months, and 12 months.

DETAILED DESCRIPTION:
OPTIMAX-OCT is a prospective, randomized (1:1), study that will be conducted at 2-3 sites (Finland, Belgium) to evaluate OPTIMAX-BAS vascular healing patterns and thrombus formation with OCT at one (Study A) and six (Study B) month after stent implantation in comparison with SYNERGY-EES. Patients receiving BAS will receive dual antiplatelet treatment (DAPT) for at least four weeks followed by aspirin, while patients implanted with EES, will receive DAPT for at least 6 months followed by aspirin.

Patients will be randomized to study A and B as follow:

Study A: OPTIMAX-BAS (n=25) versus SYNERGY-EES (n=25). First 50 patients will be randomized to study A. OCT at 1 month follow up.

Study B: OPTIMAX-BAS (n=30) versus SYNERGY-EES (n=30) Following 60 patients will be randomized to study B. OCT at 6 months follow up.

Randomization is used at the time of recruitment with sealed envelopes. Patients will be randomized in 1:1 fashion. First 50 patients are randomized in study A and following 60 patients in study B. Patients in study A will have OCT follow up at 1 month after index procedure and patients in study B will have OCT at 6 months.

OCT analyses will be performed blinded to patient's characteristics as well as the type of the stent used.

Two (2-3) investigational sites:

* Cardiovascular Center Aalst, Aalst, Belgium
* Heart Center, Satakunta Central Hospital, Pori, Finland

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <80 years
2. STEMI or NSTEMI (assumed by investigator to be type 1 myocardial infarction, according to universal definitions of MI; EHJ 2007; 28(20):2525-38); or unstable angina (clinical symptoms of chest pain, ecg suggestive of reversible ischemia)
3. Patient is willing to comply with specified follow-up evaluations
4. Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics committee or Institutional Review Board.
5. Single de novo or non-stented restenosis lesion
6. Patients with two-vessel disease may have undergone successful treatment of the non-target vessel with approved devices up to and including the index procedure but must be prior to the index target vessel treatment.
7. Target lesion (maximum 20 mm length by visual estimation) to be covered by a single stent of maximum 23mm length.
8. Reference vessel diameter must be >2.5mm and <4.0mm by visual estimate.
9. The vessel diameter should be measured after pre-dilation procedure and after intracoronary nitroglycerin if vasospasm is suspected.
10. Target lesion >50% and <100% stenosed by visual estimate.

Exclusion Criteria:

1. Impaired renal function (serum creatinine >177micromol/l) or on dialysis
2. Platelet count < 10 e5 cells/mm3
3. Patient has a history of bleeding diathesis or coagulopathy or patients in whom antiplatelet and and/or anticoagulation therapy is contraindicated.
4. Patient has received organ transplant or is on a waiting list for any organ transplant.
5. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/prasugrel/ticagrelol, cobalt chromium alloy, or contrast agent that cannot be adequately pre-medicated.
6. Patient presents with cardiogenic shock.
7. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study.
8. Currently participating in another investigational drug or device study.
9. Unprotected left main disease.
10. Ostial target lesions.
11. Chronic total occlusion.
12. Calcified target lesions that cannot be adequately pre-dilated.
13. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment.
14. Target lesion involving bifurcation with a side branch larger than 2.0mm in diameter.
15. A >30% stenosis proximal or distal to the target lesion that cannot be covered with the same stent.
16. Diffuse distal disease.
17. Prior stent in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the percentage of stent struts coverage per group | 1 month
  In Study A, time for the OCT primary endpoint is 1month
Primary endpoint is the percentage of stent struts coverage per group | 6 months
  In Study B, time for the OCT primary endpoint is 6 month

SECONDARY OUTCOMES:
Percentage of stent strut malapposition | 1 and 6 months
Maximum length of segment (mm) with uncovered stent struts | 1 and 6 months
Maximum length of segment (mm) with malapposed stent struts | 1 and 6 months
Maximum malapposition distance | 1 and 6 months
Total malapposition volume | 1 and 6 months
Mean neointimal thickness | 1 and 6 months
Percentage of protruding struts per stent | 1 and 6 months
Stent area | 1 and 6 months
NIH volume | 1 and 6 months
Thrombus formation | 1 and 6 months
In-stent late loss | 6 months
In-segment late loss | 6 months
In-stent binary restenosis | 6 months
In-segment binary restenosis | 6 months
Major adverse cardiac events defined as a composite of death, MI (Q wave or non-Q wave), emergent coronary artery bypass surgery (CABG), or justified target lesion revascularization (TLR) | 1, 6, and 12 months
Target vessel revascularization | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pasi P Karjalainen, MD, phd, Study Director — Heart Center, Satakunta Central Hospital
Locations (2):
- Cardiovascular Center Aalst, OLV-Clinic, Aalst, Belgium, Aalst, Belgium
- Heart Center, Satakunta Central Hospital, Pori, Finland

REFERENCES:
- [Derived] Sia J, Nammas W, Collet C, De Bruyne B, Karjalainen PP. Comparative study of neointimal coverage between titanium-nitric oxide-coated and everolimus-eluting stents in acute coronary syndromes. Rev Esp Cardiol (Engl Ed). 2023 Mar;76(3):150-156. doi: 10.1016/j.rec.2022.05.017. Epub 2022 Jun 2. English, Spanish. PMID 35752571